CLINICAL TRIAL: NCT06959836
Title: Post-market Safety and Performance Outcomes of the VIVERE® Bovine Pericardial Bioprosthetic Valve
Acronym: VITTA
Status: Completed | Type: Observational
Sponsor: Braile Biomedica Ind. Com. e Repr. Ltda. (Industry)
Responsible Party: Sponsor
Other Study IDs: VITTA
Record Dates: First submitted 2025-04-23; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: AORTIC VALVE DISEASES; Aortic Valve Stenosis and Insufficiency; Aortic Valve Surgery; Mitral Valve Regurgitation; Mitral Valve Surgery
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis; Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: VIVERE Bovine Pericardial Bioprosthetic Valve — Replacement of the native valve or bioprosthesis

SUMMARY:
This study aims to collect post-market safety and performance data related to the procedure and follow-up of the VIVERE Bovine Pericardial Bioprosthetic Valve, when used in accordance with the product's Instructions for Use (IFU).

DETAILED DESCRIPTION:
A multicenter, observational, retrospective, single-arm study. This study will include patients who underwent valve replacement (native or bioprosthetic) of the aortic or mitral valves using the VIVERE Bovine Pericardial Bioprosthetic Valve, between 2017 and 2022. Data will be collected up to 3 years post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* All patients who received the VIVERE® Bovine Pericardial Bioprosthetic Valve for replacement of the native valve or bioprosthesis in the aortic or mitral position, in accordance with the Instructions for Use (IFU).
* Patients aged > 18 years.

Exclusion Criteria:

* Patients who received the VIVERE® Bovine Pericardial Bioprosthetic Valve for replacement of the tricuspid or pulmonary valve.
* Contraindications specified in the IFUs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent aortic or mitral valve replacement (native valve or bioprosthesis) with the VIVERE® Bovine Pericardial Bioprosthetic Valve.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Safety performance | Hospital discharge or within 30 days of the procedure, whichever occurs first.
  Procedure- or device-related mortality
Efficacy outcome | 3 years post-implant
  Percentage of patients in NYHA (New York Heart Association functional classification) Class I or II at 3 years post-implant.

SECONDARY OUTCOMES:
Clinical success | Hospital discharge
  Defined as valve implantation without complications and without serious adverse events up to hospital discharge
Composite serious valve-related adverse events (non-linearized) | From immediately after the intervention until study completion, with an average follow-up of 3 years
  Defined as death, stroke, and/or reintervention within 3 years of valve implantation
Hemodynamic Performance | From immediately after the intervention until study completion, with an average follow-up of 3 years
  Effective orifice area (cm²), mean pressure gradient (mmHg) and paravalvular leak.
Structural Valve Deterioration | 30 days, 1 year, 2 years, and 3 years
  Defined as calcification, fibrosis, and/or leaflet fracture.
Serious Adverse Events (linearized rates) | 30 days, 1 year, 2 years, and 3 years
  Bleeding, thromboembolism, valve thrombosis (thrombus formation with prosthetic dysfunction), endocarditis (infection leading to prosthetic dysfunction), non-structural valve dysfunction (leak, mismatch, and/or late embolization), and structural valve deterioration (calcification, fibrosis, and/or leaflet fracture), paravalvular leak, need for reintervention, and valve-related or non-valve-related death.
All-Cause Mortality | 3 years post-valve implantation
  Including cardiovascular and non-cardiovascular causes, within 3 years after implantation.

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Hospital Nossa Senhora (Fundação Pio Xii), Barretos, São Paulo
  - Hospital de Caridade São Vicente de Paulo, Jundiaí, São Paulo
  - Hospital Beneficência Portuguesa, São José do Rio Preto, São Paulo

IPD SHARING:
Plan to Share IPD: No